CLINICAL TRIAL: NCT05512078
Title: Assessment of Vertical Ridge Augmentation for Posterior Mandible Using Computer Guided Onlay Versus Free Hand Onlay Grafting Procedures: A Randomized Clinical Split Mouth Trial
Brief Title: Assessment of Vertical Ridge Augmentation for Posterior Mandible by Computer Guided Onlay vs Free Hand Onlay Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamid Khorshed, principle investigator, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: omf10721
Record Dates: First submitted 2022-07-23; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Vertical Deficeny of Posterior Mandible
Keywords: vertical posterior mandible

STUDY DESIGN:
Intervention Model Description: patients with bilateral vertical bone loss in posterior mandible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): patient specific surgical positioning guide
  Interventions: Procedure: bone positioning surgical guide
- control (Active Comparator): onlay bone graft
  Interventions: Procedure: bone positioning surgical guide

INTERVENTIONS:
Procedure: bone positioning surgical guide — patient specific surgical positioning guide made from acrylonitrile butadiene styrene (ABS) plastic material.
  Other Names: bone fixation surgical guide

SUMMARY:
for patients with vertical bone loss in posterior mandible area......invistigators use chin blocks for vertical augmentation...i compare between using guide for positiong the block with the desired position using special surgical guide versus position the block with free hand technique

DETAILED DESCRIPTION:
• The CBCT scan images will be imported into a computer software (Mimics15, Materialise, Leuven, Belgium) for the reformatting of the retrieved DICOM images and reconstruction of three-dimensional virtual model of both the donor and recipient sites.

The virtual model will be imported into a second software (3-Matic, Materialise, Leuven, Belgium) specialized in designing medical devices and surgical stents.

* The 1st surgical guide will be designed to guide the harvesting of two bilateral bone blocks ensuring that each block is designed with the superior osteotomy line more than 5 mm away from the apices of the anterior teeth and the inferior line more than 5 mm away from the inferior border of the mandible and the medial line 5 mm away from the symphysis, with two screw holes in the symphysis area to fixate the guide to the bone.
* The 2nd surgical guide will be designed to guide the fixation of the onlay graft, the design will include two screw holes placed with minimum 2mm safety margin below the inferior alveolar canal to fixate the guide in place, and two more screw holes placed supracrestal to fixate the graft to the guide superiorly.
* Finally, the surgical guide will be printed using fused deposition modeling technology with acrylonitrile butadiene styrene (ABS) plastic material. All guides will be sterilized using 2.4% gluteraldehyde for 12 hours prior to the surgery. All surgeries will be performed by the same surgeon.

ELIGIBILITY:
Inclusion Criteria:

- Age range from 25-55 years. No sex predilection. 8

* Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
* Edentulous bilateral posterior mandible with vertically deficient alveolar ridge that is less than 7mm measured from the crest of the alveolar ridge to the inferior alveolar canal.
* Normal vertical dimension with normal inter-arch space.
* The minimum number of missing teeth in the posterior mandible alveolar ridge is two adjacent posterior teeth.

Exclusion Criteria:

* • Intra-bony lesions (e.g. cysts) or infections (e.g. abscess) that may retard the osteotomy healing.

  * Previous grafting procedures in the edentulous area

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge vertical bone height | 4months
  measuring alveolar height bone gain using cbct

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided